CLINICAL TRIAL: NCT01146275
Title: A 7-year Follow up of All Subjects Incuded in Protocol 31GB0106
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 31GB0904
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2013-11

CONDITIONS: Breast Augmentation
Keywords: Patients who participated in pilot study (31GB0601) and performed breast augmentation with previous formulation of Macrolane

ARMS (1):
- Participants in the Pilot study 31GB0601 (Other): This is an additional safety follow up 7-years post treatment, for subjects enrolled in a pilot study using a previous formulation of Macrolane for breast augmentation.
  Radiological breast examinations - MRI of breast, mammography and ultrasound of breast
  Interventions: Radiation: Radiologial breast examination

INTERVENTIONS:
Radiation: Radiologial breast examination — MRI of breast, mammography and ultrasound of breast

SUMMARY:
Several subjects included in a Pilot study (CTN 31GB0106) during 2002-2003 still had Macrolane deposits in the breast when the last study visit was performed. An additional follow up visit is planned to follow duration and safety of the former formulation of Macrolane that was used in the Pilot study (CTN 31GB0106).

DETAILED DESCRIPTION:
All subjects included in a Pilot study between 2002-2003 (CTN 31GB0106) are offered to take part in a seven year safety follow up after the initial injection of the former formulation of Macrolane into the breasts. The study will not involve any additional treatments.

The follow up will include relevant medical history, weight, breast examination, ultrasound and mammography to determine if there are/have been any safety issues since the final study visit in the Pilot study (CTN 31GB0106), as well as a comprehensive MRI investigation to assess the breast structure and determine if there are still deposits of Macrolane in the breast.

ELIGIBILITY:
Inclusion Criteria:

* Participant in 31GB0601

Exclusion Criteria:

* There are no exclusion citeria in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, MD, PhD, Principal Investigator — Akademikliniken, Stockholm
Locations (4):
- Sweden (4):
  - Akademikliniken Öresund, Malmo
  - Sophiahemmet, Stockholm
  - Akademikliniken, Stockholm
  - ProForma Clinic, Stockholm

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants in the Pilot Study 31GB0601: This is an additional safety follow up 7-years post treatment, for subjects enroled in a pilot study using a previous formulation of Macrolane for breast augmentation.
  Radiologial breast examination : MRI of breast, mammograophy and ultrasound of breast
Period: Overall Study
Arm/Group | Participants in the Pilot Study 31GB0601
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants in the Pilot Study 31GB0601
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 6

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate if the Subject Has Macrolane Deposits in the Breast Seven Years Post Treatment, Using a Comprehensive MRI Investigation
Description: The MRI investigation was performed to evaluate if the subjects has study product (Macrolane-a Hyaluronic acid) in their breast 7 years after the treatment.
Time Frame: 7 years +/- 6months post treatment
Population: MRI were performed by 4 women out of 6. One woman was pregnant and therefore not included and one did not want to perform MRI.
Measure: Number; unit: participants with remaining product
Groups:
- Participants in the Pilot Study 31GB0601: This is an additional safety follow up 7-years post treatment, for subjects enrolled in a pilot study using a previous formulation of Macrolane (Hyaluronic acid) for breast augmentation.
  Radiologial breast examination : MRI of breast, mammography and ultrasound of breast The MRI investigation was performed to evaluate if the subjects has study product (Macrolane-a Hyaluronic acid) in their breast 7 years after the treatment.
Arm/Group | Participants in the Pilot Study 31GB0601
Number analyzed (Participants) | 4
participants with remaining product | 4

2. Primary Outcome: To Evaluate the Long Term Safety of Macrolane in Breast Enhancement
Description: To evaluate the long term safety of Macrolane in breast enhancement, using relevant medical history, breast examination, mammography and ultrasound as well as a comprehensive MRI investigation.
  Participants with AE/SAE since participation in study 31GB0106 or any findings at the breast examination, mammography, ultrasound or comprehensive MRI investigation
Time Frame: 7 years +/- 6 months post treatment
Population: Subjects that participated in study 31GB0106 was asked to partícipate in the study 31GB0904. 6 subjects signed Informed consent for this study.
Measure: Number; unit: participants
Groups:
- Participants in the Pilot Study 31GB0601: This is an additional safety follow up 7-years post treatment, for subjects enrolled in a pilot study using a previous formulation of Macrolane (Hyaluronic acid) for breast augmentation.
  Participants with AE/SAE since participation in study 31GB0106 or any findings at the breast examination, mammography, ultrasound or comprehensive MRI investigation
Arm/Group | Participants in the Pilot Study 31GB0601
Number analyzed (Participants) | 6
participants | 0

ADVERSE EVENTS:
Groups:
- Participants in the Pilot Study 31GB0601: This is an additional safety follow up 7-years post treatment, for subjects enrolled in a pilot study using a previous formulation of Macrolane for breast augmentation.
  Radiologial breast examination : MRI of breast, mammograophy and ultrasound of breast
Arm/Group | Participants in the Pilot Study 31GB0601
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less